CLINICAL TRIAL: NCT06703775
Title: Low Level Laser Versus Neural Mobilization of Brachial Plexus on Shoulder Dysfunction Post Liver Donation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hayam Abd Elrazek Mohamed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005253
Record Dates: First submitted 2024-11-20; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low level laser therapy (LLLT) + Conventional physical therapy program (Experimental): This group will be composed of 22 patients with shoulder dysfunction post liver donation. Patients will receive low level laser in addition to conventional physical therapy program. LLLT will be applied for 3 times a week for 4 consecutive weeks.
  Interventions: Other: Low level laser therapy (LLLT); Other: Conventional physical therapy program
- Neural mobilization techniques + Conventional physical therapy program (Experimental): This group will be composed of 22 patients with shoulder dysfunction post liver donation. Patients will receive neural mobilization techniques in addition to conventional physical therapy program. Exercises will be applied for 3 times a week for 4 consecutive weeks.
  Interventions: Other: Neural mobilization techniques; Other: Conventional physical therapy program
- Conventional physical therapy program (Active Comparator): This group will be composed of 22 patients with shoulder dysfunction post liver donation. Patients will receive conventional physical therapy program. Exercises will be applied for 3 times a week for 4 consecutive weeks.
  Interventions: Other: Conventional physical therapy program

INTERVENTIONS:
Other: Low level laser therapy (LLLT) — The first experimental will receive LLLT using the Fisioline Lumix 2 (Italy). Participants will be placed in a comfortable, supported sitting position and will wear protective eyeglasses to prevent retinal damage. The LLLT (GaAs type, 1-10 mW, 904 nm) will be applied to the most painful points on the deltoid and/or upper trapezius muscles. Treatment will target a minimum of two and a maximum of four painful points, with each point irradiated for 3-4 minutes, for a total session duration of up to 15 minutes.
  Arms: Low level laser therapy (LLLT) + Conventional physical therapy program
Other: Neural mobilization techniques — The second experimental will receive Neural Mobilization Therapy (NMT). The procedure will begin by positioning the patient in a sitting position. The initial positioning will involve placing the patient's arm at their side with the elbow bent at 90 degrees. The therapist will gently extend the patient's shoulder (moving the arm backward) while keeping the elbow bent, creating tension on the axillary nerve. This tension will be held for a few seconds, ensuring it remains within the patient's tolerance and does not cause discomfort or pain. The shoulder will then be slowly returned to the initial position, releasing the tension on the nerve. This sequence of tension and release will be repeated, gradually increasing the range of motion as tolerated. The treatment will consist of three sets of 10 repetitions, with a one-minute rest between sets, performed three times per week for a total of 12 sessions over four weeks.
  Arms: Neural mobilization techniques + Conventional physical therapy program
Other: Conventional physical therapy program — The following exercises will be performed by the patients of three groups. Pendulum exercise, Isometric Scapular Retraction, Rotator cuff exercise, Wall creeping exercise, Active assisted ROM exercises, Codman exercises. Each exercise will be performed for all movements namely flexion extension and abduction-adduction, one sets of each 10-15 repetitions within pain-free range and instructed to carry out their activities of daily living.

SUMMARY:
The purpose of the study will be to compare therapeutic effect of low level laser versus neural mobilization techniques on shoulder dysfunction post liver donation.

DETAILED DESCRIPTION:
The need for this study develops from the lack of information in the published studies about the effectiveness of low level laser and neural mobilization of brachial plexus on shoulder dysfunction post liver donation.

Following liver donation and transplantation, shoulder dysfunction and discomfort occur in 20% to 60% of patients.

Low-level laser therapy (LLLT) has been used as a non-pharmacological alternative to treat painful musculoskeletal conditions. It is used in acute, chronic painful and inflammatory affections shows that low energy irradiation from lasers alters cellular processes, producing anti-inflammatory effects and increased collagen turnover.

Neural mobilization (NM) is an intervention aimed at restoring the homeostasis in and around the nervous system, by mobilization of the nervous system itself or the structures that surround the nervous system. Neural mobilization facilitates movement between neural structures and their surroundings (interface) through manual techniques or exercise. Human and animal studies revealed that NM reduces intraneural edema, improves intraneural fluid dispersion, reduces thermal and mechanical hyperalgesia and reverses the increased immune responses.

The present study is designed to investigate the effect of LLLT versus NMT on shoulder dysfunction post liver donation.

ELIGIBILITY:
Inclusion Criteria:

* Patients are both males and females.
* Their age will range from (20-50) years.
* Patients will suffer from unilateral shoulder pain(Rt shoulder).
* Patients will begin the training program one week post.operative.
* All patients will suffer from moderate to severe pain (VAS score > 4).
* Patients will be given their informed consent.

Exclusion Criteria:

* Known history of high level Spinal cord injury and malignancy
* Metabolic disease with a neurological component such as diabetes.
* Orthopedic disorders such as fracture or dislocation.
* Musculoskeletal disorders that will impair performance during training and tests.
* Uncontrolled cardiovascular or pulmonary diseases .
* Circulatory disturbances of upper extremity
* Psychiatric illness, severe behavior or cognitive disorders.
* Uncooperative patients.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-11-26 (Estimated); Primary Completion 2025-01-26 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Arabic version of Shoulder Pain and Disability Index (SPADI) | 4 weeks
  The SPADI is a self-reported questionnaire with 13 items divided into two subscales: pain and disability. The pain subscale includes five questions about pain intensity during specific activities, such as lying on the involved side, reaching for a high shelf, or pushing with the involved arm. The disability subscale has eight questions about difficulty with tasks like washing hair, putting on clothing, or carrying a 10-pound object. Each question is rated on an 11-point scale (0-10). Scores are summed, converted to percentages, and averaged to provide a total SPADI score ranging from 0 (best) to 100 (worst). SPADI will be assessed pre- and post-treatment (4 weeks).

SECONDARY OUTCOMES:
Measurement of shoulder flexion range of motion (ROM) | 4 weeks
  It will be measured from supine lying position, using a digital goniometer. The starting position for the participant's arm will be beside his body with the elbow extended and the thumb pointing upward. The axis of measurement will be the lateral part of greater tubercle and the lateral epi-condyle as the reference point. The fixed arm will be placed parallel to the surface of the floor, the movable arm will be placed parallel to the lateral aspect of the upper arm (humerus).
Measurement of shoulder abduction range of motion (ROM) | 4 weeks
  It will be measured from supine lying position, using a digital goniometer. The starting position for the participant's arm will be laterally rotated beside his body with the elbow extended and palm facing upward without flexion or extension of shoulder. The axis of measurement will be the anterior aspect of the acromion process and the medial epicondyle as the reference point. The fixed arm will be placed parallel to the surface of the floor, the movable arm will be placed parallel to the anterior aspect of the upper arm (humerus).
Measurement of shoulder external rotation range of motion (ROM) | 4 weeks
  It will be measured from supine lying position, using a digital goniometer. The starting position for the participant's arm was abducted 900 and elbow flexed 90° with the forearm perpendicular on the plinth, with his palm facing toward his feet without forearm pronation or supination and elbow outside plinth, a small pad was used under the humerus to be in level with the acromion. The distal end of humerus, thorax, and clavicle was stabilized. The axis of measurement was the olecranon process, and the ulnar styloid process as the reference point.
Measurement of maximum isometric force (MIF) of shoulder abductors | 4 weeks
  The maximum isometric force (MIF) of shoulder abductors will be measured before and after treatment period using Lafayette hand-held dynamometer. The MIF will be measured through an accommodating isometric "make" test, where participants applied maximal force against the examiner while a steady position was maintained. Participants will perform three, 5 seconds contractions for each muscle group with a 30 second rest after each trial and 5 minutes rest between muscle groups. The average force of the three testing trials will be computed for each muscle. The examiner encourages participants to do their best effort during measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Mohamed Abd El-baky, PhD, Study Chair — Professor, Cairo university
Locations (1):
- faculty of physical therapy, Cairo University, Giza, Egypt